CLINICAL TRIAL: NCT02392663
Title: Sputum Clearance Effects of Hypertonic Saline in Non-cystic Fibrosis Bronchiectasis: a Randomized, Double-blind, Crossover Trial
Brief Title: Sputum Clearance Effects of Hypertonic Saline in Non-cystic Fibrosis Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Eva Polverino, Post doctoral investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Hyperosmolar_NCFB
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Bronchiectasis
Keywords: Sputum clearance; Cough severity; Hypertonic saline; Acid hyaluronic; Tolerability
MeSH Terms: conditions — Bronchiectasis | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hypertonic saline solution (Active Comparator): Hypertonic saline (7%) solution (5 ml) will be nebulized by all patients in a randomized order. Immediately after, patients will perform a bronchial drainage session. The airway clearance technique selected will be autogenic drainage (AD).
  Both patients and physiotherapist will be blind to the intervention.
  Interventions: Other: Hypertonic saline solution
- Hyaneb solution (Active Comparator): Hyaneb (acid hyaluronic + hypertonic saline [7%]) solution (5 ml) will be nebulized by all patients in a randomized order. Immediately after, patients will perform a bronchial drainage session. The airway clearance technique selected will be autogenic drainage (AD).
  Both patients and physiotherapist will be blind to the intervention.
  Interventions: Other: Hyaneb solution
- Isotonic saline solution (Placebo Comparator): Isotonic saline (0,9%) solution (5 ml) will be nebulized by all patients in a randomized order. Immediately after, patients will perform a bronchial drainage session. The airway clearance technique selected will be autogenic drainage (AD).
  Both patients and physiotherapist will be blind to the intervention.
  Interventions: Other: Isotonic saline solution

INTERVENTIONS:
Other: Hypertonic saline solution — All patients will perform 4 sessions during the same week. Each session will be include: inhalation period + bronchial drainage period. 20 minutes will be spent to perform the inhalation period. Moreover, 30 minutes will be spent to complete the bronchial drainage session post-inhalation.
  Arms: Hypertonic saline solution
Other: Hyaneb solution — All patients will perform 4 sessions during the same week. Each session will be include: inhalation period + bronchial drainage period. 20 minutes will be spent to perform the inhalation period. Moreover, 30 minutes will be spent to complete the bronchial drainage session post-inhalation.
  Arms: Hyaneb solution
Other: Isotonic saline solution — All patients will perform 4 sessions during the same week. Each session will be include: inhalation period + bronchial drainage period. 20 minutes will be spent to perform the inhalation period. Moreover, 30 minutes will be spent to complete the bronchial drainage session post-inhalation.
  Arms: Isotonic saline solution

SUMMARY:
This study aims to analyze whether the hypertonic saline nebulization enhances sputum clearance effects, reduces the impact on cough severity and their level of safety and tolerability in a population with non-cystic fibrosis bronchiectasis (NCFBE). In addition, this trial aims to compare these health outcomes among 3 nebulized solutions: hypertonic saline (7%); hyaluronic acid + hypertonic saline (7%); isotonic saline (0,9%).

DETAILED DESCRIPTION:
The present study will be a randomized, double-blind, crossover trial. Each nebulized solution [hypertonic saline (7%); hyaluronic acid + hypertonic saline (7%); isotonic saline (0,9%)] will be administrated during 4 days. After each inhalation, all patients will carry out a bronchial drainage session (autogenic drainage technique). All patients recruited will perform the three arms of intervention. In this way, each patient will be able to act as his/her own control.

A 7 days washout period will be required among the different solutions to avoid carryover effects.

During the study period the patients' pharmacological treatment remained unchanged.

ELIGIBILITY:
Inclusion Criteria:

1. Non-cystic Fibrosis bronchiectasis (NCFBE) diagnosed by High Resolution Computed Tomographic
2. Mean sputum production ≥ 10 ml /24h.
3. Clinical stability in the last 4 weeks
4. To be able to understand how to perform inhalation and the physiotherapy session.
5. To be able to provide written, informed consent

Exclusion Criteria:

1. Forced expiratory volume in 1 second < 30% pred. ; Total lung capacity < 45% pred.
2. Performing nebulization with any hyperosmolar agents, previously
3. Allergic bronchopulmonary aspergillosis diagnosis
4. Not to be able to overcome the safety test pre-intervention (oxygen saturation levels drop to < 90% and/or forced expiratory volume in 1 second decline more than < 12% from baseline during the nebulization process)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Wet sputum production | 1h wet sputum production (g)
  Sputum collected during nebulization period and physiotherapy session

SECONDARY OUTCOMES:
Wet sputum production | 24h wet sputum production (g)
  Spontaneous sputum expectorated during the following 24h after intervention
Impact on cough severity (Leicester Cough Questionnaire) | One week
  Self-administered questionnaire (Leicester Cough Questionnaire)
Lung function (Forced spirometry) | One week
  Forced spirometry: forced expiratory volume in 1 second, Forced vital capacity, Forced expiratory flow 25-75
Safety and tolerability (Adverse events) | 20 minutes
  Adverse events registration during the nebulization process (heart rate, saturation and dyspnoea)

OTHER OUTCOMES:
Patients´preference (Likert test) | 5 weeks
  Self-administered "Likert test" at the end of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Eva Polverino, Dr., Principal Investigator — Hospital Clinic
Locations (1):
- Hospital Clinic, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Herrero-Cortina B, Alcaraz-Serrano V, Torres A, Polverino E. Reliability and Minimum Important Difference of Sputum Weight in Bronchiectasis. Respir Care. 2020 Oct;65(10):1478-1487. doi: 10.4187/respcare.07175. Epub 2020 Feb 18. PMID 32071136